CLINICAL TRIAL: NCT00064779
Title: Pilot Imaging Study to Assess the Distribution of IL13-PE38QQR Cytotoxin Infusions in Patients With Recurrent, Resectable, Supratentorial Malignant Glioma
Brief Title: Imaging Study of the Distribution of IL13-PE38QQR Infused Before and After Surgery in Adult Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IL13PEI-105
Record Dates: First submitted 2003-07-11; First posted 2003-07-15 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Malignant Glioma; Glioblastoma Multiforme; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Mixed Oligoastrocytoma
Keywords: CNS neoplasms; Brain neoplasms; neurosurgery; intralesional infusion; recombinant proteins; immunotoxins
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma; Oligodendroglioma; Central Nervous System Neoplasms; Brain Neoplasms | interventions — IL13-PE38; Surgical Procedures, Operative

INTERVENTIONS:
Drug: IL13-PE38QQR
Procedure: targeted fusion protein therapy
Procedure: surgery

SUMMARY:
The experimental anti-cancer drug IL13-PE38QQR, which is being developed for the treatment of malignant brain tumors, is composed of parts of two proteins: the immune system cytokine IL13 and a toxin from the bacterium Pseudomonas aeruginosa. The IL13 part of the drug binds to another protein, the IL13 receptor, when this receptor is displayed on the outside surface of cells. Cells with drug bound to the IL13 receptor take up the drug, and the toxin part of the drug then kills those cells. Since brain tumor cells display the IL13 receptor, they are potential targets that may be killed by this drug. This is a pilot study to visualize the distribution of IL13-PE38QQR infused into and around brain tumor tissue before and after surgical removal of the tumor in adult patients with recurrent malignant glioma.

Stored tumor tissue will be tested for presence of the receptor protein, which is required for study entry. Eligible patients will then undergo biopsy to confirm the diagnosis of recurrent malignant glioma. IL13-PE38QQR will be infused for 96 hours into and around tumor tissue through catheters that have been placed surgically. For the first 48 hours the drug will be mixed with a radioactive tracer, so that the distribution of the drug can be followed by a type of scanning called SPECT. Surgery to remove the tumor will be performed approximately 15 days after the end of the infusion. Catheters will again be placed surgically, and IL13-PE38QQR will be infused a second time for 96 hours. Radioactive tracer will be included in the infusion for the first 48 hours. For both infusions, SPECT scans will be taken at 6, 24, and 48 hours after the start of infusion. MRI scans will be taken within 90 minutes of the 24 and 48 hour SPECT scans. Patients will be followed closely with further scans and laboratory tests until completion of the study approximately 58 days after completion of the second infusion.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the distribution of IL13-PE38QQR following continuous infusion via catheter(s) into recurrent malignant glioma prior to surgical resection and a continuous infusion via catheter(s) into brain tissue adjacent to tumor resection site after surgical resection. 123I-HSA tracer will be used as a surrogate for study drug distribution.
* Determine the toxicities associated with administration of IL13-PE38QQR as described above.
* Assess the effect on distribution of IL13-PE38QQR of varying the catheter type (up to 3) and flow rate per catheter, keeping the total flow rates constant, for the pre- and post-resection infusions.

OUTLINE: This is a pilot study to assess the distribution of IL13-PE38QQR delivered by intratumoral infusion prior to surgical resection and by interstitial infusion into tissue surrounding the resection site (peritumoral) after surgical resection. Prior to resection, catheters will be placed in the region of the solid contrast-enhancing tumor component. The volume of infusion, the duration of infusion, and the concentration of IL13-PE38QQR in the infusate will be fixed. For the post-resection infusion, catheters will be placed peritumorally into areas at greatest risk for residual or infiltrating tumor. The post-resection volume of infusion, the duration of infusion, and the concentration of IL13-PE38QQR in the infusate will be fixed. For the first 48 hours of each infusion, IL13-PE38QQR will be prepared with 123I-HSA tracer as the surrogate for distribution of study drug. The type and number of catheters utilized to deliver the pre- and post-surgery infusions will vary. To maintain a fixed total volume of infusate over 96 hours, the rate of infusion will vary depending upon the number of catheters utilized. Up to three different catheter types will be tested. However, only the same, single type of catheter will be utilized for the pre- and post-resection infusions for a given patient.

To allow assessment of the distribution of the infused material, the first 48 hours of both the pre- and post-resection infusions will utilize 123I-HSA in the infusate. For the last 48 hours of both infusions, the 123I-HSA will be replaced by non-labeled HSA. The distribution of the 123I-HSA tracer will be measured by Single-Photon Emission Computed Tomography (SPECT) scanning.

PROJECTED ACCRUAL: Up to 18 patients will be enrolled at a single site.

ELIGIBILITY:
DISEASE CHARACTERISTICS

* Archival tumor sample must express IL13Rα2 by immuno-histochemistry (IHC) analysis
* Must have prior histologic diagnosis of supratentorial malignant glioma (Grade 3 or 4), including glioblastoma multiforme, anaplastic astrocytoma, anaplastic oligodendroglioma, or mixed oligoastrocytoma (excludes glioma of unknown grade). Patients with clinical/radiographic diagnosis of malignant glioma may be registered pending histologic confirmation.
* Must have undergone prior surgical resection and received external beam radiotherapy with at least 48 Gy tumor dose, completed at least 8 weeks prior to study
* Must have recurrent or progressive supratentorial malignant glioma compared with a previous diagnostic study
* Baseline tumor measured within 2 weeks prior to study entry
* Stereotactic biopsy at study entry must confirm the presence of glioma (malignant, unless previously documented)
* Recurrent or progressive tumor must have a solid contrast-enhancing region at least 1.0 cm and no more than 5.0 cm in maximum diameter. One satellite lesion is permitted if separated by 3 cm or less from the primary mass.

PATIENT CHARACTERISTICS

* Age 18 and over
* Karnofsky Performance Score of at least 70
* Absolute neutrophil count at least 1500/mm^3
* Hemoglobin at least 10 gm/dL
* Platelet count at least 100,000/mm^3
* PT and aPTT within institutional limit of normal
* Must be candidate for re-operation
* Must have recovered from toxicity of prior therapy. Minimum intervals required: at least 6 months after approved intratumoral chemotherapy (e.g. carmustine wafer), at least 6 weeks after nitrosourea-containing chemotherapy, at least 4 weeks after any investigational agent or any other cytotoxic chemotherapy, at least 2 weeks after vincristine or non-cytotoxic chemotherapy
* Must practice an effective method of birth control during the study
* Must understand the investigational nature of this study and its potential risks and benefits, and sign an approved written informed consent prior to performance of any study-specific procedure
* No patients with tumor crossing the midline (tumor involving corpus callosum is permitted if not crossing midline), more than two foci of tumor, or non-parenchymal tumor dissemination (e.g. subependymal or leptomeningeal)
* No patients with impending herniation (e.g. midline shift greater than 1.0 cm), uncontrolled seizures, or requirement for immediate palliative treatment
* No patients who have received localized therapy for glioma, e.g. focal single-fraction radiotherapy, brachytherapy, or intracerebral infusion of chemotherapy or cytotoxin
* No patients who are receiving any concurrent chemotherapy or any other investigational agent (corticosteroids are permitted)
* No patients with a known allergy to iodine or to contrast medium that may be utilized in scans required by this protocol
* Female patients must not be pregnant or breast-feeding
* No patients unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2003-07; Primary Completion 2006-06 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States